CLINICAL TRIAL: NCT03580876
Title: Addition of Azathioprine to the Switch of Anti-TNF Drug in IBD Patients in Clinical Relapse With Undectectable Anti-TNF Trough Levels and Anti-drug Antibodies : a Prospective Randomized Trial
Brief Title: Addition of Azathioprine in IBD Patients With Immunogenic Failure
Acronym: Comboswitch
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Védrines, Philippe, M.D. (Individual)
Responsible Party: Principal Investigator, Philippe VEDRINES, head of gastroenterology unit and principal investigator, Védrines, Philippe, M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMBOSWITCH
Record Dates: First submitted 2018-06-12; First posted 2018-07-09 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Clinical Failure After Switch

STUDY DESIGN:
Intervention Model Description: two strategies
Masking Description: open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- switch to anti-TNF alone (Other): Switch to the second anti-TNF drug alone (infliximab or adalimumab)
  Loss of response under Infliximab: 10 mg/kg IV every 8 weeks Randomization to: Adalimumab: induction 160/80 mg SC and Maintenance 40 mg EOW SC OR Loss of response under Adalimumab: 40mg EW SC Randomization to: Infliximab: 5mg/kg IV at W0, W2, W6 and every 8 weeks.
  Interventions: Drug: Switch to a second anti-TNF drug alone
- switch to anti-TNF with addition of azathioprine (Other): Switch to anti-TNF (infliximab or adalimumab) with addition of azathioprine
  Loss of response under Infliximab: 10 mg/kg IV every 8 weeks Randomization to: Adalimumab: induction 160/80 mg SC and Maintenance 40 mg EOW SC with azathioprine 2.5 mg/kg/day OR
  Loss of response under Adalimumab: 40mg EW SC Randomization to:
  Infliximab: 5mg/kg IV at W0, W2, W6 and every 8 weeks with azathioprine 2.5 mg/kg/day.
  Interventions: Drug: addition of azathioprine

INTERVENTIONS:
Drug: addition of azathioprine — impact of addition of azathioprine after a switch of a second anti-TNF agent
  Arms: switch to anti-TNF with addition of azathioprine
Drug: Switch to a second anti-TNF drug alone — Switch to a second anti-TNF drug alone without addition of azathioprine
  Arms: switch to anti-TNF alone

SUMMARY:
Loss of response under anti-TNF is frequent. 20% of patients with clinical relapse present an immune mediated pharmacokinetic failure. In the last AGA recommendations, switch to another anti-TNF drug is suggested with no indication of immunosuppressive agent. In a recent study, 70% of patients with an immunogenic failure to a first anti-TNF agent developed a new immunogenic failure to the second anti-TNF drug using alone.

DETAILED DESCRIPTION:
The aim of the study in these patients with an immune mediated pharmacokinetic failure was to compare two strategies:

Switch to a second anti-TNF alone or switch to a second anti-TNF with addition of azathioprine

Comparing rates of clinical failure, rates of immunogenic failure and finally adverse events during a follow-up of 24 months

ELIGIBILITY:
Inclusion Criteria:

* IBD Patients in clinical failure under anti-TNF (Infliximab (IFX) or Adalimumab (ADA) in monotherapy at the optimal dose) ADA: 40mg/7 days, IFX: 10mg/kg/8 weeks Active disease CD: HBI > 5 with Calprotectin > 250 µg/g stool UC: Total Mayo Score > 4 with an endoscopic subscore > 1 Anti-TNF monotherapy for at least 4 months and optimization for at least two months
* Patients with an immune mediated PK failure Undetectable rates of anti-TNF and high Ab against anti-TNFs > 20ng/mL for ATI and AAA (Elisa Theradiag) on two consecutive samples
* Patients who have agreed to and signed the consent form

Exclusion Criteria:

* Unclassified colitis
* Pregnant woman
* Crohn's disease CD with a exclusive anoperineal phenotype
* Contraindication or intolerance to azathioprine
* Primary non-responder patients To the first anti-TNF or After the switch to a - second anti-TNF
* Ostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-07-23 (Estimated); Primary Completion 2019-06-10 (Estimated); Study Completion 2020-06-10 (Estimated)

PRIMARY OUTCOMES:
clinical failure | 24 months
  clinical relapse or serious adverse event requiring stopping treatment during follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic of Montbrison, Montbrison, Pays de la Loire Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Patton PH, Timmer A. Azathioprine and 6-mercaptopurine for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD000478. doi: 10.1002/14651858.CD000478.pub5. PMID 40013523